CLINICAL TRIAL: NCT00818142
Title: Support Group Surveys for Individuals Who Have Type 1 Diabetes and an Eating Disorder
Status: Completed | Type: Observational
Sponsor: HealthPartners Institute (Other)
Collaborators: International Diabetes Center at Park Nicollet (Other); Park Nicollet Eating Disorder Institute (Other); Park Nicollet Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 03653-07-A
Record Dates: First submitted 2009-01-05; First posted 2009-01-07 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2013-08

CONDITIONS: Eating Disorder; Type 1 Diabetes
MeSH Terms: conditions — Feeding and Eating Disorders; Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- eating disorder, type 1 diabetes: Individuals diagnosed with type 1 diabetes and an eating disorder who withhold their insulin.
  Interventions: Behavioral: ED/DM Support Group

INTERVENTIONS:
Behavioral: ED/DM Support Group — The ED/DM Recovery Group focuses on assisting individuals with diabetes and an eating disorder - specifically the struggle of withholding insulin. The group utilizes strategies and tools that have been taught in other EDI programs, and also builds on the strengths of a group. The group is a means for learning and support as the individuals continue a regular schedule of school, work, and/or family life.

SUMMARY:
We propose to conduct a monthly group of persons with type 1 diabetes who also withhold insulin. Subjects will be asked to complete a 2-page survey (check-in sheet) at the beginning of each session and a 5-page survey (Diabetes and Eating Disorders Survey) on their first session and at their last session of their group.

ELIGIBILITY:
Inclusion Criteria:

* Have an eating disorder
* Have type 1 diabetes
* Withhold their insulin
* 18 years or older
* Actively being treated at EDI
* Committed to at least one appointment each month with each member of their individual EDI team (RD, CDE or RN, CDE; LP; and MD)
* Approval of participation by EDI/DM team (RD; RN; LP; MD)
* Able to attend 66% of group sessions

Exclusion Criteria:

* Psychologically not ready for this group therapy
* Have additional eating disorder issues that would make attendance in this group inappropriate
* Not committed to continuing treatment at PN's EDI
* Not being actively treated at PN's EDI
* Has type 2 diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals diagnosed with type 1 diabetes and an eating disorder who manipulate their insulin will be considered to join the ED/DM Recovery Group.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2008-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Adherence to insulin regimen. | Monthly

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Powers, PhD, RD, CDE, Principal Investigator — International Diabetes Center at Park Nicollet
Locations (1):
- Park Nicollet Eating Disorder Institute, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Colton P, Olmsted M, Daneman D, Rydall A, Rodin G. Disturbed eating behavior and eating disorders in preteen and early teenage girls with type 1 diabetes: a case-controlled study. Diabetes Care. 2004 Jul;27(7):1654-9. doi: 10.2337/diacare.27.7.1654. PMID 15220242
- [Background] Goebel-Fabbri AE, Fikkan J, Connell A, Vangsness L, Anderson BJ. Identification and treatment of eating disorders in women with type 1 diabetes mellitus. Treat Endocrinol. 2002;1(3):155-62. doi: 10.2165/00024677-200201030-00003. PMID 15799208